CLINICAL TRIAL: NCT06355960
Title: Effect of Different Does of Dexmedetomidine on Oxygenation and Lung Mechanics
Brief Title: Effect of Dexmedetomidine on Oxygenation and Lung Mechanics
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Samir Wahdan, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-853
Record Dates: First submitted 2024-03-28; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Drug Use; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Active Comparator): Dexmedetomidine (Precedex) loadings of 1 μg/kg than continuously at a rate of 0.2 μg/(kg/h) till the end of the operation .
  Interventions: Drug: GROUP Dexmedetomidine
- group B (Active Comparator): Dexmedetomidine (Precedex) loadings of 0.5 μg/kg then continuously at a rate of 0.2 μg/(kg/h) till the end of the operation .
  Interventions: Drug: GROUP B
- group C (Active Comparator): Dexmedetomidine (Precedex) loadings of 0.25 μg/kg(group C) then continuously at a rate of 0.2 μg/(kg/h) till the end of the operation .
  Interventions: Drug: GROUP C

INTERVENTIONS:
Drug: GROUP Dexmedetomidine — Dexmedetomidine (Precedex) loadings of 1 μg/kg , then continuously at a rate of 0.2 μg/(kg/h) till the end of the operation .
  Arms: group A
Drug: GROUP B — Dexmedetomidine (Precedex) loadings of 0.5 μg/kg , then continuously at a rate of 0.2 μg/(kg/h) till the end of the operation .
  Arms: group B
Drug: GROUP C — Dexmedetomidine (Precedex) loadings of 0.25 μg/kg, then continuously at a rate of 0.2 μg/(kg/h) till the end of the operation .
  Arms: group C

SUMMARY:
Dexmedetomidine is a selective α -2 agonist widely used in anesthesia for its sympatholytic, sedative and analgesic effects . Favorable respiratory effects in animals , and in selected human patient groups have been reported when using this agent .we investigated the effects of different doses of dexmedetomidine infusion on oxygenation

ELIGIBILITY:
Inclusion Criteria:

Morbidly obese patients with restrictive lung disease ASA I AND II laparoscopic sleeve gastrectomy

Exclusion Criteria:

history of heart failure history of cardiac arrhythmias severe liver or kidney impairment. Patients with forced expiratory volume in 1 sec (FEV1)/ FVC < 70%

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Oxygenation by the end study | UP TO 6 HOURE
  PaO2/Fraction of inspired oxygen

SECONDARY OUTCOMES:
Intraoperative dynamic lung compliance | up to 6 hours
  tidal volume/ (peak airway pressure -PEEP)
Intraoperative static lung compliance | UP TO 6 HOURE
  Tidal volume/ (plateau pressure - PEEP)
Physiological dead space | UP TO 6HOURE
  1.14 (PaCO2-EtCO2)/ PaCO2-0.005

CONTACTS AND LOCATIONS:
Overall Officials: Amr s wahdan, MD, Principal Investigator — Cairo university , Cairo, Egypt
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
still working